CLINICAL TRIAL: NCT06007677
Title: A Phase 2 Long-Term Open-Label Trial to Assess the Safety and Efficacy of Repeat Dosing of STAR-0215 in Adult Patients With Hereditary Angioedema (The ALPHA-SOLAR Trial)
Brief Title: A Long-term Study of STAR-0215 in Participants With Hereditary Angioedema
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Astria Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAR-0215-202; 2023-506540-16 (EudraCT Number)
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Hereditary Angioedema
Keywords: HAE; Angioedema; Long-term; Safety
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Regimen 1 (Arm A): STAR-0215 (Experimental): Participants will receive STAR-0215 every 3 months.
  Interventions: Drug: STAR-0215
- Dose Regimen 2 (Arm B): STAR-0215 (Experimental): Participants will receive STAR-0215 every 6 months.
  Interventions: Drug: STAR-0215
- Dose Regimen 1 (Arm C): STAR-0215 (Experimental): STAR-0215 will be administered as a subcutaneous injection.
  Interventions: Drug: STAR-0215
- Dose Regimen 3 (Arm D): STAR-0215 (Experimental): STAR-0215 will be administered as a subcutaneous injection.
  Interventions: Drug: STAR-0215

INTERVENTIONS:
Drug: STAR-0215 — STAR-0215 will be administered as a subcutaneous injection.

SUMMARY:
The goal of this trial is to enable the collection of information about long-term safety and clinical activity of STAR-0215 in participants with hereditary angioedema (HAE). Participants will receive repeat doses of STAR-0215 for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Open to participants from STAR-0215-201 (NCT05695248) who have met one of the following conditions:

  * Completed STAR-0215-201 (follow up through 6 months after their last dose);
  * Eligible for STAR-0215-201 and entered the Run-In period but did not qualify for the Treatment Period because they did not meet the criterion for the minimum number of HAE attacks;
  * Eligible for STAR-0215-201 and entered the Run-In period but did not complete it for reasons other than not meeting the criterion for the minimum number of HAE attacks (eligibility requires consultation with the Medical Monitor); or
  * Discontinued STAR-0215-201 (for reasons other than safety) after having completed at least 84 days of trial follow-up since their last dose of STAR-0215 (eligibility requires consultation with the Medical Monitor).
* Open to participants who are STAR-0215 naïve and were not enrolled in STAR-0215-201 (NCT05695248), have a documented diagnosis of HAE (Type 1 or Type 2).

Exclusion Criteria:

* Any concomitant diagnosis of another form of chronic angioedema, such as acquired C1 inhibitor deficiency, HAE with normal C1-esterase inhibitor protein (also known as HAE Type III), idiopathic angioedema, or angioedema associated with urticaria.
* Any exposure to angiotensin-converting enzyme inhibitors or any estrogen-containing medications with systemic absorption (such as hormonal contraceptives or hormone replacement therapy) within 28 days prior to Screening
* Any exposure to androgens (for example, stanozolol, danazol, oxandrolone, methyltestosterone, testosterone) within 7 days prior to Screening.
* Use of therapies prescribed for the prevention of HAE attacks prior to Screening:

  * lanadelumab within 90 days
  * berotralstat within 21 days
  * all other prophylactic therapies, discuss with the Medical Monitor

Note: Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Treatment-emergent Adverse Events | Day 1 through study completion, an average of 6 years

SECONDARY OUTCOMES:
Change From Baseline in Monthly HAE Attack Rate | Day 1, up to 5 years
Severity of HAE Attacks Experienced by Participants | Day 1 through up to 5 years
  All HAE attacks will be classified according to severity (mild, moderate, and severe).
Duration of HAE Attacks | Day 1 through up to 5 years
  Duration will be reported as shorter than 12 hours, 12 to 24 hours, 24 to 48 hours, and longer than 48 hours.
Number of Participants Experiencing HAE Attacks Requiring On-demand Therapy | Day 1 through up to 5 years
Time to First HAE Attack After Each Dose | Day 1 through up to 5 years
Number of HAE Attack-free Days | Day 1 through up to 5 years
Number of Participants Experiencing Zero HAE Attacks | Day 1 through up to 5 years
Serum Concentration of STAR-0215 | Every 3 months for first 2 years, Every 6 months for next 3 years
  Blood samples will be collected on dosing days to measure the serum concentration of STAR-0215.
Plasma Levels of Cleaved High-molecular-weight Kininogen | Every 3 months for first 2 years, Every 6 months for next 3 years
  Blood samples will be collected on dosing days to measure the plasma levels of cleaved high-molecular-weight kininogen (a measure of plasma kallikrein activity).
Number of Participants with Anti-drug Antibodies to STAR-0215 | Every 3 months for first 2 years, Every 6 months for next 3 years
  Blood samples will be collected on dosing days to assess the formation of STAR-0215 anti-drug antibodies in serum.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (12):
  - Allervie Clinical Research, Birmingham, Alabama
  - Medical Research of Arizona a Division of Allergy, Asthma & Immunology Associates, LTD, Scottsdale, Arizona
  - Acuro Research, Little Rock, Arkansas
  - UC San Diego US HAEA Angioedema Center, San Diego, California
  - Raffi Tachdjian MD, Inc, Santa Monica, California
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - Institute for Asthma and Allergy, PC, Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Optimed Research, Columbus, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas
- Diagnostic Consultative Center Convex Ltd., Sofia, Bulgaria
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Ottawa Allergy Research Corporation, Ottawa, Ontario
- Institute of Clinical Immunology/Allergology, Faculty Hospital, Hradec Kralove, Hradec Králové, Czechia
- Germany (3):
  - Charité Universitätsmedizin Berlin, Berlin
  - Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt
  - Universitätsklinikum Ulm, Ulm
- Szpital Uniwersytecki w Krakowie, Krakow, Poland
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge
  - St. James's Hospital, Leeds

IPD SHARING:
Plan to Share IPD: No